CLINICAL TRIAL: NCT02029040
Title: A Randomized Trial of Nebulized 3% Hypertonic Saline in the Treatment of Acute Bronchiolitis in The Emergency Department
Brief Title: Nebulized 3% Hypertonic Saline in the Treatment of Acute Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU 012013-040
Record Dates: First submitted 2014-01-03; First posted 2014-01-07 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Acute Bronchiolitis
Keywords: Bronchiolitis; Hypertonic saline; Emergency Department
MeSH Terms: conditions — Bronchiolitis; Emergencies | interventions — Saline Solution, Hypertonic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3% hypertonic saline group (Experimental): Once consented, the study drug (in this arm: 3% Hypertonic Saline) will be ordered by a physician at the request of a study team member. Once the drug order set is received by a pharmacist, he/she will obtain the study drug from an Omnicell and prepare the medication to a volume of 3 mL in a syringe with a blinded study label prepared in advance by the IDS pharmacy. The pharmacist will then give the study drug to the patient's respiratory therapist or the bedside nurse. The respiratory therapist or the nurse will pour the drug from a syringe to an inhaler cup and the study drug will be given by the standard nebulizer over the course of 15 minutes.
  Interventions: Drug: 3% Hypertonic Saline
- 0.9% normal saline group (Placebo Comparator): Once consented, the study drug (in this arm: 0.9% normal saline) will be ordered by a physician at the request of a study team member. Once the drug order set is received by a pharmacist, he/she will obtain the study drug from an Omnicell and prepare the medication to a volume of 3 mL in a syringe with a blinded study label prepared in advance by the IDS pharmacy. The pharmacist will then give the study drug to the patient's respiratory therapist or the bedside nurse. The respiratory therapist or the nurse will pour the drug from a syringe to an inhaler cup and the study drug will be given by the standard nebulizer over the course of 15 minutes.
  Interventions: Drug: 0.9 % normal saline

INTERVENTIONS:
Drug: 3% Hypertonic Saline — Within 5-15 minutes following the administration of the study drug, the Respiratory Distress Assessment Instrument (RDAI) score will be reassessed and study interventions are complete. The patient will be observed for one hour in the emergency department (ED). However, further treatments may be started immediately upon discretion of the treating physician. If the patient is discharged home study PI and/or research assistant will call the parents 7 days from the ED visit to check the number of visits to their primary doctor and/or EDs due to same illness.
  Other Names: Experimental
  Arms: 3% hypertonic saline group
Drug: 0.9 % normal saline — Within 5-15 minutes following the administration of the study drug, the Respiratory Distress Assessment Instrument (RDAI) score will be reassessed and study interventions are complete. The patient will be observed for one hour in the emergency department (ED). However, further treatments may be started immediately upon discretion of the treating physician. If the patient is discharged home study PI and/or research assistant will call the parents 7 days from the ED visit to check the number of visits to their primary doctor and/or EDs due to same illness.
  Other Names: Placebo
  Arms: 0.9% normal saline group

SUMMARY:
This is a randomized, double-blind, controlled trial in the Pediatric Emergency Department. The primary objective is to determine whether nebulized 3% hypertonic saline is more effective than nebulized 0.9% saline in the treatment of bronchiolitis in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Children 2-12 months of age presenting to Emergency Department
* Patients with a diagnosis of bronchiolitis defined as the first episode of wheezing and/or crackles in a child younger than 12 months who has physical findings of a viral respiratory infection and has no other explanation for the wheezing and/or crackles
* Patients with an RDAI score ≥ 6 as measured by a trained respiratory therapist

Exclusion Criteria:

* Previous history of wheezing
* Known heart or lung disease
* Premature birth defined as birth before 37 weeks gestation
* Immunosuppression or immunodeficiency
* Treatment with corticosteroids in the previous 48 hours
* Critically ill children - progressive respiratory failure requiring higher level of care, vital signs instability/need for emergency interventions to prevent clinical deterioration
* Oxygen saturation <85% on room air at the time of recruitment

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Badawy, MD, Study Director — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center; Children's Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.9% Normal Saline Group; Hypertonic Saline Group: Once consented, the study drug (in this arm: 0.9% normal saline) will be ordered by a physician at the request of a study team member. Once the drug order set is received by a pharmacist, he/she will obtain the study drug from an Omnicell and prepare the medication to a volume of 3 mL in a syringe with a blinded study label prepared in advance by the IDS pharmacy. The pharmacist will then give the study drug to the patient's respiratory therapist or the bedside nurse. The respiratory therapist or the nurse will pour the drug from a syringe to an inhaler cup and the study drug will be given by the standard nebulizer over the course of 15 minutes.
  3% Hypertonic Saline versus 0.9 % normal saline: Within 5-15 minutes following the administration of the study drug, the Respiratory Distress Assessment Instrument (RDAI) score will be reassessed and study interventions are complete. The patient will be observed for one hour in the emergency department (ED).
Period: Overall Study
Arm/Group | 0.9% Normal Saline Group | Hypertonic Saline Group
Started | 27 | 25
Completed | 27 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 3% Hypertonic Saline Group: Once consented, the study drug (in this arm: 3% Hypertonic Saline) will be ordered by a physician at the request of a study team member. Once the drug order set is received by a pharmacist, he/she will obtain the study drug from an Omnicell and prepare the medication to a volume of 3 mL in a syringe with a blinded study label prepared in advance by the IDS pharmacy. The pharmacist will then give the study drug to the patient's respiratory therapist or the bedside nurse. The respiratory therapist or the nurse will pour the drug from a syringe to an inhaler cup and the study drug will be given by the standard nebulizer over the course of 15 minutes.
  Within 5-15 minutes following the administration of the study drug, the Respiratory Distress Assessment Instrument (RDAI) score will be reassessed and study interventions are complete. The patient will be observed for one hour in the emergency department (ED). However, further treatments m
- 0.9% Normal Saline Group: Once consented, the study drug (in this arm: 0.9% normal saline) will be ordered by a physician at the request of a study team member. Once the drug order set is received by a pharmacist, he/she will obtain the study drug from an Omnicell and prepare the medication to a volume of 3 mL in a syringe with a blinded study label prepared in advance by the IDS pharmacy. The pharmacist will then give the study drug to the patient's respiratory therapist or the bedside nurse. The respiratory therapist or the nurse will pour the drug from a syringe to an inhaler cup and the study drug will be given by the standard nebulizer over the course of 15 minutes.
  Within 5-15 minutes following the administration of the study drug, the Respiratory Distress Assessment Instrument (RDAI) score will be reassessed and study interventions are complete. The patient will be observed for one hour in the emergency department (ED). However, further treatments may
- Total: Total of all reporting groups
Arm/Group | 3% Hypertonic Saline Group | 0.9% Normal Saline Group | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 27 | 52
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 9.8 (6.3) | 9.2 (5.4) | 9.6 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 18 | 17 | 35
Region of Enrollment [Number; unit: participants]
  United States | 25 | 27 | 52

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Assessment Change Score (RACS)
Description: The primary outcome variable is the Respiratory Assessment Change Score (RACS) which is a sum of the change in the Respiratory Distress Assessment Instrument (RDAI)score plus a standardized score for the change in respiratory rate; the change in respiratory rate is assigned 1 point per each 10% change in the respiratory rate.The RDAI score is the sum of the row scores, with total range 0 to 17; higher scores indicate more severe disease.
Time Frame: 5-15 minutes
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 3% Hypertonic Saline Group | 0.9% Normal Saline Group
Number analyzed (Participants) | 10 | 15
score on a scale | 1.68 [0.52 to 2.84] | 1.70 [0.70 to 2.70]

2. Secondary Outcome: Rate of Hospitalizations
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | 3% Hypertonic Saline Group | 0.9% Normal Saline Group
Number analyzed (Participants) | 25 | 27
participants | 9 | 11

ADVERSE EVENTS:
Groups:
- 3% Hypertonic Saline Group: Once consented, the study drug (in this arm: 3% Hypertonic Saline) will be ordered by a physician at the request of a study team member. Once the drug order set is received by a pharmacist, he/she will obtain the study drug from an Omnicell and prepare the medication to a volume of 3 mL in a syringe with a blinded study label prepared in advance by the IDS pharmacy. The pharmacist will then give the study drug to the patient's respiratory therapist or the bedside nurse. The respiratory therapist or the nurse will pour the drug from a syringe to an inhaler cup and the study drug will be given by the standard nebulizer over the course of 15 minutes.
  Within 5-15 minutes following the administration of the study drug, the Respiratory Distress Assessment Instrument (RDAI) score will be reassessed and study interventions are complete.
- 0.9% Normal Saline Group: Once consented, the study drug (in this arm: 0.9% normal saline) will be ordered by a physician at the request of a study team member. Once the drug order set is received by a pharmacist, he/she will obtain the study drug from an Omnicell and prepare the medication to a volume of 3 mL in a syringe with a blinded study label prepared in advance by the IDS pharmacy. The pharmacist will then give the study drug to the patient's respiratory therapist or the bedside nurse. The respiratory therapist or the nurse will pour the drug from a syringe to an inhaler cup and the study drug will be given by the standard nebulizer over the course of 15 minutes.
  Within 5-15 minutes following the administration of the study drug, the Respiratory Distress Assessment Instrument (RDAI) score will be reassessed and study interventions are complete.
Arm/Group | 3% Hypertonic Saline Group | 0.9% Normal Saline Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 0/25 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes